CLINICAL TRIAL: NCT02664506
Title: Theory-Driven Treatment of Language and Cognitive Processes in Aphasia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of Pennsylvania (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Nadine Martin, Nadine Martin, Ph.D., Temple University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21987; 5R01DC013196 (NIH)
Record Dates: First submitted 2016-01-15; First posted 2016-01-27 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Word repetition after a tiem delay (Experimental): People with Aphasia and Short-Term Memory impairment will receive a behavioral treatment: Word repetition after a time delay. This is the intervention: repetition of words after a 5 or 10 second delay.
  Interventions: Behavioral: Word repetition after a time delay.

INTERVENTIONS:
Behavioral: Word repetition after a time delay. — This is a behavioral intervention, Word repetition after a time delay. Individuals listen to words and repeat them after 5 or 10 seconds.
  Other Names: Repetition after delay

SUMMARY:
The aim of this research is to translate a theory of the cognitive relationship between verbal short--term memory (STM) and word processing impairments in aphasia to treatment approaches for language impairment in aphasia. It has been proposed that the co-occurrence of these impairments is due to a disruption of cognitive processes that support both abilities: maintenance of activated semantic and phonological representations of words, hereafter the 'activation--maintenance hypothesis'.

This hypothesis will be tested in the context of a treatment approach that aims to improve word processing and verbal STM abilities. The grant supporting this work has ended. therefore, participants are entered into the study by invitation only.

DETAILED DESCRIPTION:
Based on research of word processing and verbal STM impairments in aphasia, it has been proposed that the co-occurrence of these impairments is due to a disruption of cognitive processes that support both abilities: maintenance of activated semantic and phonological representations of words, hereafter the 'activation--maintenance hypothesis'.

This hypothesis will be tested in the context of a treatment approach that aims to improve word processing and verbal STM abilities. Recently, the importance of treatment research has been emphasized as a critical testing ground for theories of language processing. Although it has been demonstrated that associations between impairments of word processing and reduced verbal STM capacity support the 'activation-maintenance hypothesis', direct treatments to improve the ability to maintain activation of word representations will serve as a stronger test of this hypothesis. First, empirical support will be established for the hypothesis that impairment to short-term maintenance of activated semantic and phonological representations of words impairs language and verbal STM abilities in aphasia and that direct treatment of this deficit will improve both abilities (Specific Aim 1). Second, the effects of this treatment will be compared under two administration conditions, high and low intensity (Specific aim 2). Finally, the neural regions associated with semantic STM and phonological STM will be investigated using voxel--based lesion--symptom mapping (Bates et al., 2003) (Specific Aim 3).

This research represents a unique attempt to apply more recent processing theories of aphasia to treatment of the disorder.The outcomes will have important implications for aphasia rehabilitation research.

ELIGIBILITY:
Experimental participants:

Inclusion Criteria:

* Aphasia
* Single left hemisphere lesions
* Right handed
* At least six months post-stroke
* Aged 21 to 80
* High-school educated with English as their primary language
* Passed an audiometric pure tone, air conduction screening at 25 dB HL at 1K, 2K and 4K Hz for at least one ear (with or without correction)
* Demonstrate adequate vision with or without correction.
* Will not exclude individuals with a mild apraxia of speech or mild dysarthria of speech.

Exclusion Criteria:

* History of mental illness
* Alcohol/substance abuse
* Pregnant
* Unable to personally give informed consent

Control participants:

Inclusion Criteria:

* Aged 21 to 80
* High school educated or above
* Pass an audiometric pure tone, air conduction screening at 25 dB HL at 1K, 2K and 4K Hz for at least one ear.

Exclusion Criteria:

* History of neurological disease or language disability
* Histories for mental illness
* Alcohol/substance abuse.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Verbal Short-Term Memory (STM) Span at 6 weeks | Baseline and 6 weeks
  It is expected that this treatment will increase verbal STM span (primary)

SECONDARY OUTCOMES:
Change in proportion of words retrieved in picture naming | Post treatment, after 6 weeks of treatment
  More words will be retrieved accurately in picture naming.
Discourse measures, changes in rates of context information units | Post treatment, after 6 weeks of treatment
  Proportion of content information units will increase as a consequence of htis therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Martin, Ph.D., Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No